CLINICAL TRIAL: NCT04257773
Title: International REACH Forgiveness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: Harvard University (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Dr. HO Man Yee, Assistant Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CityUHK
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Mental Health Wellness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants in this group will receive treatment/intervention immediately.
  Interventions: Behavioral: REACH Forgiveness Workbook Intervention
- Delayed Treatment (Experimental): Participant in this group will receive treatment/intervention 2-week later.
  Interventions: Behavioral: REACH Forgiveness Workbook Intervention

INTERVENTIONS:
Behavioral: REACH Forgiveness Workbook Intervention — Participants will be asked to complete the REACH Forgiveness Workbook

SUMMARY:
Six sites spanning five regions (Hong Kong, Colombia, Indonesia, Ukraine, South Africa) will administer a forgiveness workbook intervention in a randomized design with a stepped, waitlist intervention deployment.

DETAILED DESCRIPTION:
Intervention deployment:

ODO1 X O2 O3 (immediate-treatment [IT ] group) ODO1 O2 X O3 (delayed-treatment [DT ] group)

where OD denotes measurement of baseline demographic and personality measures, X denotes deployment of the intervention, and O1, O2, and O3 denote measurements of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and comprehend the materials in the workbook
* Must be 18 years old or above
* Have someone in mind they want to forgive

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4598 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Depression (BSI) | 4 months
  Brief Symptom Index, minimum value = 0, maximum value = 4. Higher scores indicates a higher psychological distress.
Anxiety (BSI) | 4 months
  Brief Symptom Index. minimum value = 0, maximum value = 4. Higher scores indicates a higher psychological distress.
Forgiveness (TRIM) | 4 months
  Transgression-Related Interpersonal Motivations, minimum value = 1, maximum value = 5. The higher the score, the more unforgiving the person is.

SECONDARY OUTCOMES:
Trait Forgiveness (TSF) | 4 months
  Trait Forgiveness Scale, minimum value = 1, maximum value = 5. The higher the whole score, the more forgiveness the person is.
Forbearance (FS) | 4 months
  Forbearance Scale, minimum value = 1, maximum value = 6. The higher the score, the higher forbearing the person is.
Decision to Forgive (DTSF) | 4 months
  Decision to Forgive Scale, minimum value = 1, maximum value = 5. The higher the score, the higher decisional forgiveness of the subject.
Flourishing | 4 months
  Flourishing Index, minimum value = 1, maximum value = 10. The higher the score, the higher flourishing of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Man Yee Ho, PhD, Principal Investigator — City University of Hong Kong
Locations (5):
- Universidad del Sinú, Córdoba, Colombia
- Universitas Gunadarma, Depok, Indonesia
- The South African and Africa Chapter of the International Association of Assessing Officers, Pretoria, South Africa
- Ukraine (2):
  - Realis Center for Education and Research, Kyiv
  - Ukrainian Institute of Arts and Sciences, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Data, which will be used for meta-analysis, reproducibility, and replication purposes, will be disclosed after the embargo period (30 April, 2024).
Supporting Information: Study Protocol, Analytic Code
Time Frame: After the embargo period (30 April, 2024)

REFERENCES:
- [Derived] Ho MY, Worthington EL, Cowden RG, Bechara AO, Chen ZJ, Gunatirin EY, Joynt S, Khalanskyi VV, Korzhov H, Kurniati NMT, Rodriguez N, Anastasiya Salnykova A, Shtanko L, Tymchenko S, Voytenko VL, Zulkaida A, Mathur MB, VanderWeele TJ. International REACH forgiveness intervention: a multisite randomised controlled trial. BMJ Public Health. 2024 Mar 13;2(1):e000072. doi: 10.1136/bmjph-2023-000072. eCollection 2024 Jun. PMID 40018096